CLINICAL TRIAL: NCT03446300
Title: The Cohort Study of Early Visual Impairment Mechanism Caused by Change of Fundus Structure in Adults With High Myopia
Brief Title: Shanghai High Myopia Study for Adults
Acronym: SHMSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Other Study IDs: YFZX2018002
Record Dates: First submitted 2018-02-10; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: High Myopia
Keywords: High Myopia, fundus structure, early visual impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- college student population
- working population
- aged more than 50 years old population

SUMMARY:
High myopia retinopathy has become the first cause of irreversible blindness and severe visual impairment in Chinese adults, in order to avoid the blind and visual impairment caused by high myopia retinopathy, it is very necessary to research the mechanism of early visual impairment to prevent and control damages. Our recent research found that the decreasing of macular retina vascular density and subfoveal choroidal thickness, the increasing of Beta Zone area in optic atrophy and the rising of glycosylated hemoglobin in high myopia patients were significantly related to visual impairment, which suggested that the source of visual impairment was the abnormal structure changes surrounding optic and fovea, but so far there is no related study. We will conduct a 5 years prospective cohort study in the population of 2420 high myopia and controls which have established in college student population, working population and aged more than 50 years old population, using the latest OCT-A and SS-OCT to measure macular retina vascular density, subfoveal choroidal thickness, Beta Zone area in optic atrophy, combined with the semiparametric mixed effects model, we will analysis the prediction index between fundus structure parameters, blood biochemical index and individual characteristics prediction to explore the public health management mode of early prevention and treatment during high myopia population.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old; spherical equivalent refraction ≤-6.00D;

Exclusion Criteria:

* a history of ocular or systemic diseases including congenital cataract and glaucoma; previous intraocular or refractive surgery;other evidence of retinal pathology

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: college student population; working population; aged more than 50 years old population.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Retina Vessel Density (RVD) | December 31, 2016
  RVD is calculated both the macular and peripapillary area.
tilted optic disc | December 31, 2016
  A tilted optic disc was defined as the tilt ratios ≤0.80.
β-zone PPA | December 31, 2018
  The β-zone PPA area (an inner crescent of chorioretinal atrophy with good visibility of the large choroidal vessels and the sclera) was determined as the total number of pixels using the ImageJ software in a circumferential pattern.
glycosylated hemoglobin | December 31, 2020
  This test measures the average blood sugar control for the previous three months or so.

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Zhu, PhD, MD, Study Director — Shanghai Eye Disease Prevention & Treatment Center
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li M, Xu H, Ye L, Zhou S, Xie J, Liu C, Zhu J, He J, Fan Y, Xu X. Association of macular outward scleral height with axial length, macular choroidal thickness and morphologic characteristics of the optic disc in Chinese adults. Eye (Lond). 2024 Apr;38(5):923-929. doi: 10.1038/s41433-023-02804-5. Epub 2023 Oct 28. PMID 37898715